CLINICAL TRIAL: NCT02641132
Title: The Comparison of Endothelial Cell Count in Pterygium Surgery Relating to the Timing of MMC Application.
Brief Title: Pterygium Head Body MMC1: Two Different Surgical Procedures and Their Effect on Endothelial Cell Count.
Acronym: PHB-MMC1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, segev fani, Department of Ophthalmology, Meir medical centre, Kfar saba, Isreal, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0091-13-MMC
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-08

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pterygium surgery: Head and body. (Experimental): Application of Mitomycin C 0.02% after excision of the body and the head of the pterygium.
  Interventions: Drug: Mitomycin C 0.02%; Procedure: Pterygium surgery
- Pterygium surgery: Body. (Active Comparator): Application of Mitomycin C 0.02% after excision of the body only of the pterygium.
  Interventions: Drug: Mitomycin C 0.02%; Procedure: Pterygium surgery

INTERVENTIONS:
Drug: Mitomycin C 0.02% — Pterygium excision with application of mitomycin C
Procedure: Pterygium surgery — Two different procedures- excision of the head and the body and excision of the head only

SUMMARY:
To evaluate changes in endothelial cell count after pterygium surgery with mitomycin C (MMC) 0.02%

DETAILED DESCRIPTION:
To evaluate the change in endothelial cell count in patients after pterygium surgery with mitomycin C (MMC) 0.02% for 2 minutes in 2 groups.

* The control group: application of MMC after excision of the body of the pterygium without the head
* The study group: application of MMC after excision of the body and the head of the pterygium

ELIGIBILITY:
Inclusion Criteria:

* Males/females >18 Years old
* Pterygium with indication to operate
* Subjects that are able to sign an informed consent

Exclusion Criteria:

* Recurrent Pterygium/suspected tumor lesion
* Patients with endothelial cell diseases
* Patients after anterior segment surgery
* Patients with low compliance
* Patients without judgment ability
* Pregnancy
* Patients participated in another survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell count | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sackler school of medicine, Tel Aviv, Israel
  - Meir medical centre, Kfar Saba

REFERENCES:
- [Background] Avisar R, Avisar I, Bahar I, Weinberger D. Effect of mitomycin C in pterygium surgery on corneal endothelium. Cornea. 2008 Jun;27(5):559-61. doi: 10.1097/ICO.0b013e318165b158. PMID 18520505
- [Background] Bahar I, Kaiserman I, Lange AP, Slomovic A, Levinger E, Sansanayudh W, Slomovic AR. The effect of mitomycin C on corneal endothelium in pterygium surgery. Am J Ophthalmol. 2009 Mar;147(3):447-452.e1. doi: 10.1016/j.ajo.2008.08.035. Epub 2008 Nov 7. PMID 18992871
- [Background] Avisar R, Apel I, Avisar I, Weinberger D. Endothelial cell loss during pterygium surgery: importance of timing of mitomycin C application. Cornea. 2009 Sep;28(8):879-81. doi: 10.1097/ICO.0b013e3181a3900c. PMID 19654528
- [Background] Kheirkhah A, Izadi A, Kiarudi MY, Nazari R, Hashemian H, Behrouz MJ. Effects of mitomycin C on corneal endothelial cell counts in pterygium surgery: role of application location. Am J Ophthalmol. 2011 Mar;151(3):488-93. doi: 10.1016/j.ajo.2010.09.014. Epub 2011 Jan 13. PMID 21236405